CLINICAL TRIAL: NCT03841734
Title: Study of the Benefit of Early Treatment With an Endothelin Inhibitor (Bosentan) in Patients With Sudden Blindness Due to Giant Cell Arteritis: CECIBO
Acronym: CECIBO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-AOIP-01
Record Dates: First submitted 2019-02-05; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Arteritis, Giant Cell; Blindness and Low Vision
MeSH Terms: conditions — Giant Cell Arteritis; Blindness; Vision, Low | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment bosentan (Experimental)
  Interventions: Drug: treatment

INTERVENTIONS:
Drug: treatment — 8 patients will be treat with bosentan at 145 mg per day during 14 days

SUMMARY:
Giant cell arteritis , also named Horton's disease, is the most common vasculitis in subjects over 50 years old. The incidence increases with age : from 188 to 290 cases per million inhabitants per year, with a North-South gradient.

The major risk of Horton's disease is blindness, unilateral, occurring in 15 to 20% of cases, sometimes preceded by episodes of transient amaurosis. The decrease in visual acuity is often brutal, irreversible and bilateral in 25 to 50% of cases. The mechanism of this blindness is an arterial ischemia: Acute Anterior Ischemic Optic Neuropathy acute anterior ischaemic optic neuropathy (90%), acute retro-bulbar ischaemic optic neuropathy (5%), occlusion of the central artery of the retina (5%).

The pathogenesis of this brutal ischemia is not fully understood. One of the hypotheses suggests that, during stimulation by an antigen of the environment, preactivated dendritic cells of the arterial wall would stimulate T lymphocytes. These will recruit cells that cause an inflammatory infiltrate polymorphic predominant at the media level. These lesions may be accompanied by destruction of the internal elastic lamina, with inconstant but pathognomonic presence of multinucleated giant cells. All arteries with internal elastic lamina can be affected by parietal inflammation, which results in stenosis and occlusion, explaining the ischemia.

The visual loss is usually abrupt and very severe, leaving the patient with definitely very low or no residual visual acuity.

Conventional treatment currently recommended includes systemic corticosteroid therapy at 1 mg / kg / day, preceded or not by 500 mg pulses of methylprednisolone , and associated with antiplatelet and anticoagulant therapy (LMWH). Despite the decline in visual acuity thus occurred is then always final. Certainly loss of vision has a major impact on the quality of life of patients.

Apart from this lymphocytic inflammation, a process of vascular remodeling is at the origin of the vascular occlusion phenomenon. The endothelin system is a family of amino acids including 3 members: ET1, ET2 and ET3. ET1 is a potent vasoconstrictor. ET1 receptors (ETA and ETB) are expressed in the arteries of patients with giant cell arteritis . The expression of ET1 associated with proliferation of muscle cells in arteries will decrease under the effect of endothelin inhibitors. This has been shown during treatment of pulmonary hypertension. In giant cell arteritis , the endothelin system continues to be very active up to 8 days despite the introduction of systemic corticosteroids. Bosentan is a mixed endothelin receptor antagonist with affinity for both ETA and ETB receptors. This inhibitor is used in treatment of pulmonary artery hypertension, digital ulcerations of systemic sclerosis and critical peripheral arterial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Decreased visual acuity (BVA) <5 days, regardless of degree of severity, abrupt onset in the context of newly diagnosed or suspected Horton's disease at this loss of visual acuity
* Able to sign the consent
* Affiliated to the social security system
* Already under conventional treatment of Horton's disease or the: requiring: Corticosteroids and + - anti-platelet aggregators and / or LMWH at the discretion of the referring physician for its vasculitis and + - immunosuppressive or biotherapy if necessary.

Exclusion Criteria:

* Underlying hepatocellular insufficiency known
* Patient under guardianship or curator
* Hypersensitivity to the active substance or to any of the excipients
* Moderate to severe hepatic insufficiency corresponding to class B or C of the Child-Pugh classification
* Any other ophthalmological pathology explaining the sudden drop in vision: retinal detachment, retinal hemorrhage, posterior uveitis, nonarteritic arterial occlusion, cortical stroke
* Serum levels of hepatic aminotransferases, aspartate aminotransferases (ASTs) and / or alanine aminotransferases (ALATs), greater than 3 times the upper limit of normal before start of treatment
* Patient under treatment with cyclosporine A, antiretrovirals, glibenclamide or Rifampicin.
* Pregnant or lactating women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Visual acuity calculated according to the Early Treatment Diabetic Retinopathy Study | 3 months

SECONDARY OUTCOMES:
Visual acuity calculated according to the Early Treatment Diabetic Retinopathy Study | 1 month
Goldman's one-sided visual field | 3 months
Numbers of adverse event and serious adverse events | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Tieulié, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CH de Cannes, Cannes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaigne-Delalande S, de Menthon M, Lazaro E, Mahr A. [Giant-cell arteritis and Takayasu arteritis: epidemiological, diagnostic and treatment aspects]. Presse Med. 2012 Oct;41(10):955-65. doi: 10.1016/j.lpm.2012.07.011. Epub 2012 Aug 31. French. PMID 22940467
- [Background] Watelet B, Samson M, de Boysson H, Bienvenu B. Treatment of giant-cell arteritis, a literature review. Mod Rheumatol. 2017 Sep;27(5):747-754. doi: 10.1080/14397595.2016.1266070. Epub 2017 Jan 13. PMID 27919193
- [Background] Salvarani C, Cantini F, Hunder GG. Polymyalgia rheumatica and giant-cell arteritis. Lancet. 2008 Jul 19;372(9634):234-45. doi: 10.1016/S0140-6736(08)61077-6. PMID 18640460
- [Background] Gonzalez-Gay MA, Garcia-Porrua C, Llorca J, Hajeer AH, Branas F, Dababneh A, Gonzalez-Louzao C, Rodriguez-Gil E, Rodriguez-Ledo P, Ollier WE. Visual manifestations of giant cell arteritis. Trends and clinical spectrum in 161 patients. Medicine (Baltimore). 2000 Sep;79(5):283-92. doi: 10.1097/00005792-200009000-00001. PMID 11039076
- [Background] Weyand CM, Goronzy JJ. Medium- and large-vessel vasculitis. N Engl J Med. 2003 Jul 10;349(2):160-9. doi: 10.1056/NEJMra022694. No abstract available. PMID 12853590
- [Background] Bienvenu B, Ly KH, Lambert M, Agard C, Andre M, Benhamou Y, Bonnotte B, de Boysson H, Espitia O, Fau G, Fauchais AL, Galateau-Salle F, Haroche J, Heron E, Lapebie FX, Liozon E, Luong Nguyen LB, Magnant J, Manrique A, Matt M, de Menthon M, Mouthon L, Puechal X, Pugnet G, Quemeneur T, Regent A, Saadoun D, Samson M, Sene D, Smets P, Yelnik C, Sailler L, Mahr A; Groupe d'Etude Francais des Arterites des gros Vaisseaux, under the Aegis of the Filiere des Maladies Auto-Immunes et Auto-Inflammatoires Rares. Management of giant cell arteritis: Recommendations of the French Study Group for Large Vessel Vasculitis (GEFA). Rev Med Interne. 2016 Mar;37(3):154-65. doi: 10.1016/j.revmed.2015.12.015. Epub 2016 Jan 29. PMID 26833145
- [Background] Weyand CM, Schonberger J, Oppitz U, Hunder NN, Hicok KC, Goronzy JJ. Distinct vascular lesions in giant cell arteritis share identical T cell clonotypes. J Exp Med. 1994 Mar 1;179(3):951-60. doi: 10.1084/jem.179.3.951. PMID 8113687
- [Background] Terrades-Garcia N, Cid MC. Pathogenesis of giant-cell arteritis: how targeted therapies are influencing our understanding of the mechanisms involved. Rheumatology (Oxford). 2018 Feb 1;57(suppl_2):ii51-ii62. doi: 10.1093/rheumatology/kex423. PMID 29982777
- [Background] Lozano E, Segarra M, Corbera-Bellalta M, Garcia-Martinez A, Espigol-Frigole G, Pla-Campo A, Hernandez-Rodriguez J, Cid MC. Increased expression of the endothelin system in arterial lesions from patients with giant-cell arteritis: association between elevated plasma endothelin levels and the development of ischaemic events. Ann Rheum Dis. 2010 Feb;69(2):434-42. doi: 10.1136/ard.2008.105692. Epub 2009 Mar 15. PMID 19289383
- [Background] Dimitrijevic I, Andersson C, Rissler P, Edvinsson L. Increased tissue endothelin-1 and endothelin-B receptor expression in temporal arteries from patients with giant cell arteritis. Ophthalmology. 2010 Mar;117(3):628-36. doi: 10.1016/j.ophtha.2009.07.043. Epub 2009 Dec 24. PMID 20036012
- [Background] Planas-Rigol E, Terrades-Garcia N, Corbera-Bellalta M, Lozano E, Alba MA, Segarra M, Espigol-Frigole G, Prieto-Gonzalez S, Hernandez-Rodriguez J, Preciado S, Lavilla R, Cid MC. Endothelin-1 promotes vascular smooth muscle cell migration across the artery wall: a mechanism contributing to vascular remodelling and intimal hyperplasia in giant-cell arteritis. Ann Rheum Dis. 2017 Sep;76(9):1624-1634. doi: 10.1136/annrheumdis-2016-210792. Epub 2017 Jun 12. PMID 28606962
- [Background] Regent A, Ly KH, Groh M, Khifer C, Lofek S, Clary G, Chafey P, Baud V, Broussard C, Federici C, Labrousse F, Mesturoux L, Le Jeunne C, Vidal E, Brezin A, Witko-Sarsat V, Guillevin L, Mouthon L. Molecular analysis of vascular smooth muscle cells from patients with giant cell arteritis: Targeting endothelin-1 receptor to control proliferation. Autoimmun Rev. 2017 Apr;16(4):398-406. doi: 10.1016/j.autrev.2017.02.006. Epub 2017 Feb 14. PMID 28232168
- [Background] Matucci-Cerinic M, Denton CP, Furst DE, Mayes MD, Hsu VM, Carpentier P, Wigley FM, Black CM, Fessler BJ, Merkel PA, Pope JE, Sweiss NJ, Doyle MK, Hellmich B, Medsger TA Jr, Morganti A, Kramer F, Korn JH, Seibold JR. Bosentan treatment of digital ulcers related to systemic sclerosis: results from the RAPIDS-2 randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2011 Jan;70(1):32-8. doi: 10.1136/ard.2010.130658. Epub 2010 Aug 30. PMID 20805294
- [Background] Narvaez J, Garcia-Gomez C, Alvarez L, Santo P, Aparicio M, Pascual M, Lopez de Recalde M, Borrell H, Nolla JM. Efficacy of bosentan in patients with refractory thromboangiitis obliterans (Buerger disease): A case series and review of the literature. Medicine (Baltimore). 2016 Nov;95(48):e5511. doi: 10.1097/MD.0000000000005511. PMID 27902617
- [Result] Ly KH, Liozon E, Fauchais AL, Vidal E. [Pathophysiology of giant cell arteritis]. Rev Med Interne. 2013 Jul;34(7):392-402. doi: 10.1016/j.revmed.2013.02.037. Epub 2013 Mar 23. French. PMID 23528439